CLINICAL TRIAL: NCT01302418
Title: Testing of Respiratory Specimens for the Validation of the QIAGEN ResPlex II Advanced Panel Test and the Artus Influenza A/B RT-PCR Test
Brief Title: Collection and Testing of Respiratory Samples
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: C10-INFLUENZA-001
Record Dates: First submitted 2011-02-18; First posted 2011-02-24 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-04

CONDITIONS: QIAGEN ResPlex II Advanced Panel; Influenza A; Respiratory Syncytial Virus Infections; Infection Due to Human Parainfluenza Virus 1; Parainfluenza Type 2; Parainfluenza Type 3; Parainfluenza Type 4; Human Metapneumovirus A/B; Rhinovirus; Coxsackie Virus/Echovirus; Adenovirus Types B/C/E; Coronavirus Subtypes 229E; Coronavirus Subtype NL63; Coronavirus Subtype OC43; Coronavirus Subtype HKU1; Human Bocavirus; Artus Influenza A/B RT-PCR Test; Influenza B
Keywords: Respiratory Virus; Influenza; RSV; Parainfluenza; Metapneumovirus; Rhinovirus; Coxsackie virus; Echo virus; Adenovirus; Coronavirus; Bocavirus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Coxsackievirus Infections; Influenza, Human; Paramyxoviridae Infections; Adenoviridae Infections; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Extracted nucleic acid, Residual Universal Transport Medium
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Symptomatic: Individuals with signs and symptoms of an acute respiratory tract infection where it is suspected that such signs and symptoms are caused by a respiratory virus infection.
  Interventions: Device: artus Influenza A/B RT-PCR Test

INTERVENTIONS:
Device: artus Influenza A/B RT-PCR Test — The investigational assay, used for detecting the presence of Influenza A/B.

SUMMARY:
The study will be conducted using nasopharyngeal swab specimens collected prospectively from individuals suspected of having the signs and symptoms of an acute respiratory tract infection caused by a respiratory virus. A series of standard viral culture tests validated for routine use in the clinical laboratory, and/or a series of PCR-based Laboratory Developed Tests (PCR-LDT) validated by a central reference laboratory will be used to verify the performance of the investigational artus Influenza A/B RT-PCR test and the QIAGEN ResPlex II Advanced Panel test. From each specimen five (5) aliquots will be prepared: (a) one aliquot will be tested in real-time using the assigned viral culture reference methods; (b) one aliquot will be used to extract nucleic acid in real-time for investigational testing; (c) one aliquot of the specimen will be stored at --70C for subsequent shipment to the reference laboratory for PCR-LDT testing, (d) one aliquot will be archived at -70C for subsequent follow-up by the reference laboratory (e.g., bi-directional sequencing of positive specimens), and (e) any remaining specimen will be stored for the Fresh vs. Frozen Study. The extracted nucleic acid generated from the second aliquot (i.e., "b" above) will be split and subjected to testing by both the artus Influenza A/B RT-PCR test and the ResPlex II Advanced Panel test.

DETAILED DESCRIPTION:
Each year the morbidity and mortality associated with acute respiratory tract infections fluctuates seasonally. This rise and fall is associated with the changing prevalence of respiratory viruses in the population. Myriad respiratory viruses are responsible for these infections. For example, Influenza Virus, Respiratory Syncytial Virus (RSV), Parainfluenza Virus, Human Metapneumovirus, Rhinovirus, and Adenovirus have all been identified as causing such acute infections. Numerous pathogenic subtypes have been identified within most of these viral groups. The outbreak of Severe Acute Respiratory Syndrome (SARS) in 2003 was eventually identified as a Coronavirus; the mortality of SARS among the elderly can be as high as 50%. More recently, Human Bocavirus (HBoV) has also been identified as causing acute respiratory tract infections. In 2005 the HBoV was identified by molecular testing and was found to be the only virus identified in a subpopulation of patients suffering from respiratory tract infections. Apart from supportive measure (e.g., bed rest, hydration, etc.), there are no effective treatments for many of these viral infections; however, antiviral agents (e.g., the neuraminidase inhibitors oseltamivir or zanamivir) can be used to alleviate the severity of flu-like symptoms. Identification of a respiratory virus as the causative agent is important because it eliminates the need for treatment with antibiotics; physicians typically wait 7-10 days for symptoms to alleviate before prescribing antibiotics due to risks associated with exacerbating bacterial antibiotic resistance.

Each year the virus population fluctuates, and with it the antigenic presentation of the dominant strains that circulate through the population. Epidemics arise when larger and larger portions of the population do not have innate or acquired immunological resistance to such strain(s) in a given season. The World Health Organization (WHO) maintains a separate website dedicated to tracking outbreaks of influenza, especially avian influenza (https://www.who.int/fluvirus_tracker). These zoonotic transmissions that further adapt to enable human-to-human transmission are of the greatest concern because it is predicted that virtually all humans will be immunologically naïve. Zoonotic transmissions in the human population are monitored in the hope that a pandemic similar to the Spanish Flu of 1918 can be avoided; it is estimated that well over 25 million people died from the Spanish Flu. The United States government also maintains a separate website with resources regarding the flu and pandemic related information (http://www.pandemicflu.gov/). On June 11, 2009 the WHO raised the pandemic threat level to 6 in response to the global appearance of a new strain of swine Influenza A (subtype H1N1). The rapidity with which the H1N1 virus has spread exemplifies the notion that quickly and accurately identifying a viral pathogen associated with an outbreak is critical to global public health.

In addition to the threat of an influenza outbreak, the expansion in the number of viruses that cause acute respiratory tract infections compounds the difficulty in correctly and rapidly identifying the primary pathogen; each new virus or subtype increases the complexity of testing. Molecular diagnostic assays are ideally suited to address this complexity. Assays based on the polymerase chain reaction (PCR) can incorporate multiple primers and probes (e.g., multiplexed) in a single reaction to deal with this complexity.4 Such assays are extremely sensitive, have a high degree of specificity, and can be performed very quickly. The artus Influenza A/B RT-PCR test is a real-time PCR assay for the detection and identification of Influenza A and B, while the QIAGEN ResPlex II Advanced Panel test is a nucleic acid amplification-based assay for the detection and identification of a broad range of some of the most common respiratory viruses associated with acute respiratory tract infections. In the present study respiratory specimens will be prospectively collected and tested using the artus Influenza A/B RT-PCR test and the QIAGEN ResPlex II Advanced Panel test.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that sign the Informed Consent form required for prospectively enrolling patients into the study.
* Subjects that present at a hospital, clinic, or physician's office with the signs and symptoms of a respiratory tract infection.
* Subjects with an acute respiratory infection where said acute respiratory infection is suspected of being caused by an Influenza virus.

Exclusion Criteria:

* Subjects where the duration of the symptoms of such an acute respiratory infection is greater than or equal to 5 days (i.e., ≥5).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes individuals having the signs and symptoms of an acute respiratory tract infection suspected of being caused by a respiratory virus.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2011-02; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Arizona, Tuscon, Arizona
  - Albany Medical College, Albany, New York
  - Wadsworth Center, New York State Department of Health, Albany, New York
  - The University of North Carolina, Chapel Hill, North Carolina
  - Ohio State University, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Symptomatic
Started | 272
Completed | 254
Not Completed | 18
Not completed — Protocol Violation | 9
Not completed — Non-evaluable | 9

BASELINE CHARACTERISTICS:
Arm/Group | Symptomatic
Number analyzed (Participants) | 272
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 202
  Between 18 and 65 years | 66
  >=65 years | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126
  Male | 146
Region of Enrollment [Number; unit: participants]
  United States | 272

OUTCOME MEASURES:

1. Primary Outcome: Detection of Respiratory Viruses
Description: The presence of Influenza A or Influenza B virus.
Time Frame: Specimens will be taken within 5 days of the appearance of symptoms.
Population: All subjects meeting inclusion/ exclusion criteria and who had sufficient specimen volume.
Measure: Number; unit: participants
Arm/Group | Symptomatic
Number analyzed (Participants) | 254
participants | 83 [0.91 to 0.97]

ADVERSE EVENTS:
Time Frame: 5 months.
Arm/Group | Symptomatic
Serious Adverse Events (participants affected / at risk) | 0/272
Other Adverse Events (participants affected / at risk) | 0/272

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less